CLINICAL TRIAL: NCT06792773
Title: 2024 NewAnescat Register
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Carles Espinos Ramírez, Medical Doctor, Germans Trias i Pujol Hospital
Other Study IDs: PI-23-280
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
20 years ago, for the first time in Spain, a record was made of all the activity carried out by a medical speciality, called ANESCAT 2003. After 20 years, the increase in healthcare activity has exceeded the expectations and predictions that were made at the time. Therefore, it is necessary to make a new assessment of the work situation in which our speciality finds itself in order to be able to evaluate whether the increase in resources allocated has been proportional and therefore to be able to have objective data with a view to making new demands and planning future needs.

ELIGIBILITY:
The activity of all the areas in which the anaesthesiologist has some kind of work involvement over 24 hours during 14 days in a year is included through several questionnaires with different formats. Therefore all patients will be included without restriction criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population is all patients involving anaesthetic activity during the study days (14 days in a year).
Sampling Method: Non-Probability Sample
Enrollment: 13634 (Estimated)
Dates: Start 2025-05-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Anaesthesia surgical activity | Assessed during the 14-day cut-off period of the study over one year
  The main outcome and objective of the study is to quantify all the anaesthesia activity
Anaesthesia activity in the Intensive Care Units | Assessed during the 14-day cut-off period of the study over one year
  The main outcome and objective of the study is to quantify all the anaesthesia activity
Anaesthesia activity in the Chronic Pain Units | Assessed during the 14-day cut-off period of the study over one year
  The main outcome and objective of the study is to quantify all the anaesthesia activity
Anaesthesia activity in the delivery rooms | Assessed during the 14-day cut-off period of the study over one year
  The main outcome and objective of the study is to quantify all the anaesthesia activity

SECONDARY OUTCOMES:
Percentage of active staff in anaesthesiology services | Assessed during the 14-day cut-off period of the study over one year
  With the aim of finding out the real needs of professionals in relation to medical activity
The role of anaesthesiology services in Catalonia with regard to polytrauma patients | Assessed during the 14-day cut-off period of the study over one year
  The role of anaesthesiology services in Catalonia with regard to polytrauma patients
The role of anaesthesiology services in Catalonia with regard to cardiorespiratory arrest | Assessed during the 14-day cut-off period of the study over one year
  The role of anaesthesiology services in Catalonia with regard to cardiorespiratory arrest

CONTACTS AND LOCATIONS:
Overall Officials: Carles Espinós, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain